CLINICAL TRIAL: NCT01483703
Title: Noninvasive Optical Measurement of Critical Care Neonates
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bernard Choi, Ph.D., Assistant Professor Biomedical Engineering, University of California, Irvine
Other Study IDs: 20118163
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Signs and Symptoms
MeSH Terms: conditions — Signs and Symptoms | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic tool: Laser Speckle Imaging of Critical Care Neonates
  Interventions: Device: Laser Speckle Imaging

INTERVENTIONS:
Device: Laser Speckle Imaging — Laser Speckle Imaging of Critical Care Neonates

SUMMARY:
The purpose of this study is to determine whether reflections of light can be used to provide real-time pictures of blood vessel formation around infants' heads. This study device is called laser speckle imaging.

DETAILED DESCRIPTION:
The researchers can use the laser speckle imaging device to image superficial cerebral blood flow in the infant's head. The researchers can quantify blood flow and measured vessel diameter, versus actual diameter assessed with conventional digital camera imaging.

ELIGIBILITY:
Inclusion Criteria:

* New born or infant

Exclusion Criteria:

* non- new born or infant

Ages: 1 Minute to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Medical tool | up to 12 months
  Laser Speckle Imaging device to image superficial cerebral blood flow in the infant's head

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Choi, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- CHOC, Orange, California, United States